CLINICAL TRIAL: NCT06919289
Title: Quantifying the Phoenix Sign: A Comparative, Randomized Control Trial Analysis of Lidocaine and Papaverine-Induced Vascular Enhancement After Common Peroneal (Fibular) Nerve Blocks for the Diagnosis of a Focal Peripheral Nerve Entrapment
Brief Title: The Investigators Are Comparing Lidocaine and Papaverine Nerve Blocks to Determine Which Improves Blood Flow Better, Making the "Phoenix Sign" Clearer on Imaging. This Helps Accurately Diagnose Nerve Compression, Improving Patient Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Neuropathy Centers (Other)
Responsible Party: Principal Investigator, Stephen Barrett, US Neuropathy Centers Medical Director, US Neuropathy Centers
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Diagnostic
Other Study IDs: JIN-2025-0326; USNC-2025-3 (Other: USNC)
Record Dates: First submitted 2025-03-27; First posted 2025-04-09 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Drop Foot
Keywords: Nerve entrapment; Drop foot
MeSH Terms: conditions — Peroneal Neuropathies; Nerve Compression Syndromes

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Lidocaine group (Active Comparator): This arm is randomized to the laterality of the subject for either lidocaine or papaverine
  Interventions: Drug: Lidocaine infiltration
- Papavarine (Active Comparator): This arm is randomized to the laterality of the subject for either lidocaine or papaverine, for the first infiltration. The contralateral extremity will then receive the agent that was not administered on the first side from randomization.
  Interventions: Drug: Infiltration of papaverine

INTERVENTIONS:
Drug: Infiltration of papaverine — The study was randomized and double blinded. For randomization, the first extremity had either an infiltration of 0.5 cc of papaverine HCL (30mg/ml) for a 15mg perineural infiltration, or .5 cc of 1% lidocaine without epinephrine determined by a coin toss application.
  Arms: Papavarine
Drug: Lidocaine infiltration — The study was randomized and double blinded. For randomization, the first extremity had either an infiltration of 0.5 cc of papaverine HCL (30mg/ml) for a 15mg perineural infiltration, or .5 cc of 1% lidocaine without epinephrine determined by a coin toss application.
  Arms: Lidocaine group

SUMMARY:
This pilot study aims to investigate the effects of nerve blocks in patients with diabetic peripheral neuropathy through a double-blinded, randomized trial involving 4 patients. Each participant will receive bilateral peripheral nerve blocks using either lidocaine or papaverine. Following randomization, each patient will receive one medication in one leg and the alternate medication in the contralateral leg. Researchers will measure parameters including motor strength, sensory function (two-point discrimination), arterial blood flow via Doppler ultrasound, and microvascular perfusion using near-infrared spectroscopy both prior to and following nerve block administration. This research seeks to explore potential diagnostic and therapeutic applications for peripheral nerve entrapment, a common yet challenging clinical condition.

DETAILED DESCRIPTION:
Detailed Analysis of the Phoenix Sign and Vascular Changes Following Nerve Blocks in Diabetic Neuropathy

Study Background and Purpose

This study investigates the vascular and neurological phenomena associated with peripheral nerve blocks in patients with diabetic neuropathy. The primary aim is to assess whether observed changes following nerve block administration can be attributed to vasodilatory effects of lidocaine or neurological mechanisms.

Common peroneal nerve (CPN) entrapment is the third most common nerve entrapment pathology in humans and frequently results in foot drop, characterized by difficulty lifting the front part of the foot.

Study Design and Methodology

This pilot study is a double-blinded, randomized trial involving 4 diabetic patients presenting bilateral anterior compartment weakness affecting dorsiflexion. All participants will have confirmed diabetic neuropathy with severe sensory impairment.

Key methodological elements:

Randomized administration of 0.5 cc of papaverine HCL (30 mg/ml) or 0.5 cc of 1% lidocaine without epinephrine.

Initial randomization of the first leg via coin toss, with the contralateral leg receiving the alternate medication.

Double-blinded design, ensuring neither patients nor evaluating physicians are aware of medication allocation for each leg.

Ultrasound-guided perineural injection at the fibular neck level.

Comprehensive pre- and post-injection assessments.

Study assessments include:

Macrovascular assessment:

Ultrasound Doppler waveform analysis.

Measurement of blood flow velocity in dorsalis pedis and posterior tibial arteries.

Microvascular assessment:

Kent Snapshot Near-Infrared (NIR) imaging of dorsal and plantar foot surfaces.

Measurement of hemoglobin, deoxyhemoglobin, oxygen saturation (SpO2), and total hemoglobin.

Imaging scheduled pre-injection, at 4 minutes post-injection, and at 10 minutes post-injection.

Motor function assessment:

Movement Against Manual Resistance (MAMR) scored from 1-5 (normalized to 0.2-1.0).

Evaluation of three muscles: extensor hallucis longus (EHL), tibialis anterior (TA), and extensor digitorum longus (EDL).

Dynamometer measurements of EHL muscle strength (Newtons, N).

Sensory assessment:

Two-point discrimination testing

ELIGIBILITY:
Inclusion Criteria:

* subjects were included if they were diabetic and neuropathic.

Exclusion Criteria:

* Patients with Trypanophobia

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2024-03-07 (Actual); Primary Completion 2024-03-07 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Manual Motor Strength Testing of Anterior Compartment | From enrollment to 1 day of testing
  Movement Against Manual Resistance (MAMR) was evaluated using a scale of 1-5 out of 5. This was normalized so that 1/5 = 0.2, and 5/5=1.0. This was performed on three muscles of the anterior compartment, extensor hallusis longus (EHL), tibialis anterior (TA), and extensor digitorum longus (EDL) and the result for three muscles were averaged. In addition, the EHL was evaluated with a dynamometer, in Newtons (N) separately.

CONTACTS AND LOCATIONS:
Locations (1):
- Indiana Foot and Ankle, Jasper, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barrett SL, Boyd B, DuCasse S, Nassier W, Mitchell N, Nagra AP, Dalmau-Pastor M, Yamasaki DS, Nickerson S. Is the phoenix sign phenomenon due to vasodilation? A double-blinded, randomized controlled trial comparing motor function recovery after diagnostic common fibular nerve block with lidocaine and papaverine. BMC Musculoskelet Disord. 2024 Oct 23;25(1):840. doi: 10.1186/s12891-024-07972-3. PMID 39443927